CLINICAL TRIAL: NCT00645151
Title: A Multicenter, Eight-Week Treatment, Single Step Titration, Open-Label Study Assessing The Percentage Of Subjects Achieving Low Density Lipoprotein Cholesterol Target With Atorvastatin Starting Doses Of 10 Mg, 20 Mg, 40 Mg, And 80 Mg (Latin American Atorvastatin ATGOAL Study)
Brief Title: A Study Of The Efficacy Of Atorvastatin In Lowering Cholesterol In Latin American Patients With High Cholesterol
Acronym: LA ATGOAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581104
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Risk (Experimental)
  Interventions: Drug: Atorvastatin
- Low Risk (Experimental)
  Interventions: Drug: Atorvastatin
- Medium Risk (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin calcium 10, 20, 40, or 80 mg tablets (dose dependent on individual risk factors and baseline LDL-C level) once daily for 4 weeks. After 4 weeks of treatment, subjects who did not achieve the LDL-C target goal were up-titrated to 20, 40, or 80 mg and subjects who achieved their LDL-target goal remained on the same dose for the following 4 weeks.
  Arms: High Risk
Drug: Atorvastatin — Atorvastatin calcium 10, 20, 40, or 80 mg tablets (dose dependent on individual risk factors and baseline LDL-C level) once daily for 4 weeks. After 4 weeks of treatment, subjects who did not achieve the LDL-C target goal were up-titrated to 20, 40, or 80 mg and subjects who achieved their LDL-target goal remained on the same dose for the following 4 weeks.
  Arms: Low Risk
Drug: Atorvastatin — Atorvastatin calcium 10, 20, 40, or 80 mg tablets (dose dependent on individual risk factors and baseline LDL-C level) once daily for 4 weeks. After 4 weeks of treatment, subjects who did not achieve the LDL-C target goal were up-titrated to 20, 40, or 80 mg and subjects who achieved their LDL-target goal remained on the same dose for the following 4 weeks.
  Arms: Medium Risk

SUMMARY:
The purpose of this study is to determine the percentage of patients who would reach a cholesterol goal after atorvastatin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high cholesterol eligible for treatment with baseline LDL-C level of less than or equal to 220 mg/dL
* Willingness to follow diet

Exclusion Criteria:

* Triglycerides less than or equal to 400 mg/dL
* Hemoglobin A1c >10%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2004-04; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Responder rate in patients who achieved low-density lipoprotein cholesterol (LDL-C) level | Week 8

SECONDARY OUTCOMES:
Percentage of patients achieving LDL goal at 2 and 4 weeks | Weeks 2 and 4
Lipid changes at week 4 & 8 | Weeks 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Brazil (9):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São José, Santa Catarina
  - Pfizer Investigational Site, São Paulo, SP/Brazil
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São José do Rio Preto, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
  - Pfizer Investigational Site, Rio de Janeiro
- Pfizer Investigational Site, Santiago, Santiago Metropolitan, Chile
- Colombia (5):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bogotá, Cundinamarca
  - Pfizer Investigational Site, Barranquilla
  - Pfizer Investigational Site, Bogotá, C/marca
  - Pfizer Investigational Site, Cali, Valle
- Pfizer Investigational Site, Quito, Pichincha / Ecuador, Ecuador
- Pfizer Investigational Site, Guatemala City, Guatemala
- Mexico (5):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Chihuahua City
  - Pfizer Investigational Site, Durango
- Pfizer Investigational Site, Panama City, Panama
- Venezuela (4):
  - Pfizer Investigational Site, Caracas, Dtto Federal
  - Pfizer Investigational Site, Caracas, Edo. Miranda
  - Pfizer Investigational Site, Dtto. Federal, Miranda
  - Pfizer Investigational Site, Caracas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581104&StudyName=A%20Study%20Of%20The%20Efficacy%20Of%20Lipitor%20In%20Lowering%20Cholesterol%20In%20Latin%20American%20Patients%20With%20High%20Cholesterol